CLINICAL TRIAL: NCT04389541
Title: Clinical Research Platform on Decision Making and Clinical Impact of Biomarker-Driven Precision Oncology
Acronym: INFINITY
Status: Completed | Type: Observational
Sponsor: iOMEDICO AG (Industry)
Collaborators: Bristol-Myers Squibb (Industry); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Other Study IDs: IOM-050408
Record Dates: First submitted 2020-04-17; First posted 2020-05-15 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Advanced Solid Tumors or Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Tissue samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The retrospective cohort study INFINITY will be an instrument to analyze the current practice of precision oncology in the real-world setting. It will provide insight into real-world biomarker-directed treatment of cancer patients not eligible for standard therapies. The study will retrospectively collect medical records' data of patients who received a targeted treatment based on a potentially actionable alteration or biomarker identified by molecular diagnostics. Data of deceased patients will be included. The study will analyze how molecular test results guided clinical decision making. The compiled treatment and outcome data will be a valuable resource to analyze the use and effectiveness of targeted therapy approaches in biomarker-defined and entity-defined subpopulations of cancer patients. These signals might generate new insights and foster progress of targeted cancer treatment. The associated biomarker profiling module aims to set up a decentral biobank for future research on molecular alterations or central re-testing.

ELIGIBILITY:
Inclusion Criteria:

* Advanced solid tumors (i.e. locally advanced, inoperable and/or metastatic) or hematologic malignancies not eligible for standard therapy options (i.e. without further treatment options with drugs approved for the specific indication based on the judgement of the treating physician)
* Started or completed at the documenting study site a non-standard targeted therapy based on an actionable alteration or biomarker identified by molecular diagnostics
* Results on molecular diagnostics (e.g. tumor genomic or protein expression test) must be available; based on these results the therapy decision was taken
* Targeted therapy (given as monotherapy or as part of a therapy regimen) must be non-standard at time point of patient registration in the eCRF
* Age ≥ 18 years
* Signed and dated informed consent form (only if patient is alive at time of data entry into the project; not applicable for inclusion of deceased patients' data)

Exclusion Criteria:

* Non-standard targeted therapy was given within a clinical trial
* The targeted therapy was given in a line of treatment for which it is non-standard (e.g. treatment in first line instead of second line where it is approved); the targeted therapy is however in principle approved for the given entity
* The targeted therapy was non-standard because a certain prior treatment has not been applied (e.g. targeted therapy is only approved after platin-based treatment but has been given without prior platin-based treatment); the targeted therapy is however in principle approved for the given entity
* The targeted therapy was non-standard because a different or no chemotherapy back-bone has been applied (e.g. targeted therapy is approved in combination with cisplatin but has been given with oxaliplatin or without chemotherapy backbone); the targeted therapy is however in principle approved for the given entity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with advanced solid tumors or hematologic malignancies not eligible for standard therapies who received a targeted therapy based on an actionable alteration or biomarker identified by molecular diagnostics
Sampling Method: Non-Probability Sample
Enrollment: 499 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | Maximum 5 years
  Proportion of patients with CR or PR as best response

SECONDARY OUTCOMES:
Patient and Disease Characteristics | maximum 5 years
  Describe demographics, comorbidities and tumor type of patients not eligible for standard therapies.
Details on molecular diagnostics | Maximum 5 years
  Frequency of type of molecular diagnostic testing performed, of single gene/protein tests, multigene panels or NGS in molecular diagnostics, of type (by panel size) of NGS library sequenced, of proteins and genes tested, of altered proteins and genes, if tested, of treatment recommendations given in molecular diagnostic reports, of implemented treatment recommendations given in molecular diagnostic reports, of the use of a molecular tumor board (MTB), of implementation of the treatment recommendation given by MTB and duration from molecular testing result to start of non-standard targeted treatment
Clinical decision making | Maximum 5 years (once per targeted therapy)
  Frequency of answers rated with a Likert scale on patient's non-suitability for standard therapy options / choice of performed molecular diagnostics / choice of selected molecular target and targeted non-standard therapy / reasons for the selection of targeted non-standard therapy / primary goal of the non-standard targeted therapy / expected advantages of the non-standard targeted therapy and frequency of ESMO Scale of Clinical Actionability for molecular Targets (ESCAT) evidence levels
Evaluation of selected treatment approach assessed via project specific survey | Maximum 5 years (once per completed targeted therapy)
  Frequency of pre-defined answers on therapy duration, effectiveness and overall benefit
Best overall response | Maximum 5 years
  Proportion of patients with complete response (CR), partial response (PR), stable disease (SD) or progressive disease (PD)
Disease Control Rate | Maximum 5 years
  Proportion of patients with CR, PR or SD as best response
Time to Response | Maximum 5 years
  Time from start of treatment to the first objective tumor response (e.g., tumor shrinkage of ≥30%) observed for patients who achieved a CR or PR
Duration of Response | Maximum 5 years
  Time from documentation of tumor response to disease progression or death from any cause
Time to treatment failure | Maximum 5 years
  Time from start of therapy to discontinuation of treatment for any reason, including progression, toxicity, and death
Progression-free survival | Maximum 5 years
  Time from start of treatment until disease progression or death
PFS ratio | Maximum 5 years
  PFS ratio of targeted non-standard therapy and preceding treatment line
Overall Survival | Maximum 5 years
  Time from start of treatment until death of any cause

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Marschner, MD, Principal Investigator — Outpatient center for hematology and oncology, Freiburg, Germany
Locations (97):
- Germany (97):
  - MVZ am Klinikum Aschaffenburg, Aschaffenburg
  - Studienzentrum Aschaffenburg, Aschaffenburg
  - Onkologische Schwerpunktpraxis, Augsburg
  - Hämatologisch-Onkologische Schwerpunktpraxis Bad Liebenwerda, Bad Liebenwerda
  - Sozialstiftung Bamberg Medizinisches Versorgungszentrum am Bruderwald gemeinnützige GmbH, Bamberg
  - Onkologische Schwerpunktpraxis Bamberg, Bamberg
  - Klinikum Bayreuth; Klinik für Onkologie und Hämatologie, Bayreuth
  - Onkologisches Versorgungszentrum Friedrichshain, Berlin
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - Gemeinschaftspraxis für Onkologie und Hämatologie, Berlin
  - Evangelisches Waldkrankenhaus,Spandau,Innere Medizin I, Berlin
  - MVZ Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Onkologisch-Hämatologische Schwerpunktpraxis, Bremen
  - Klinikum Coburg Hämatologie, Onkologie, Coburg
  - Schwerpunktpraxis für Hämatologie und internistische Onkologie Coburg, Coburg
  - PIOH - Praxis Internistische Onkologie und Hämatologie, Cologne
  - Gemeinschaftspraxis für Hämatologie und Onkologie, München MVZ GmbH, Cologne
  - Klinikum Darmstadt, Onkologisches Studienzentrum, Darmstadt
  - Onkologisches Zentrum Deggendorf, Deggendorf
  - Onkozentrum Dresden/Freiberg, Dresden
  - BAG / Onkologische Gemeinschaftspraxis, Dresden
  - Onkologische Gemeinschaftspraxis, Dresden
  - MVZ Onkologie und Hämatologie am Sana Krankenhaus Gerresheim, Düsseldorf
  - Praxis und Tagesklinik für gynäkologische Onkologie, Ebersberg
  - Studienbüro CHOP GmbH, Frankfurt a.M.
  - Agaplesion Markus Krankenhaus, Frankfurt a.M.
  - Universitätsklinikum Frankfurt; Medizinische Klinik 1: Pneumologie, Gastroenterologie, Hepatologie, Frankfurt a.M.
  - Universitätsklinikum Frankfurt; Medizinische Klinik 2, Hämatologie, Onkologie, Frankfurt a.M.
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau
  - Gemeinschaftspraxis Panagiotou/Minaei (GbR), Garbsen
  - MVZ II der Niels Stensen Kliniken Onkologie u. Hämatologie, Georgsmarienhütte
  - Gemeinschaftspraxis Dres. Schmitt und Eulenbruch, Gerlingen
  - Überörtliche Berufsausübungsgemeinschaft, MVZ Onkologische Kooperation Harz, Goslar
  - OSP Göttingen Dres. Meyer / Ammon / Metz, Göttingen
  - Gemeinschaftspraxis für Innere Medizin, Hämatologie, Onkologie, Gastroenterologie, Halle
  - Hämatologisch-Onkologische Praxis Eppendorf (HOPE), Hamburg
  - Studiengesellschaft Hämato-Onkologie Hamburg Prof. Laack & Partner GbR, Hamburg
  - Hämatologisch-Onkologische Praxis Altona (HOPA), Hamburg
  - Onkologische Schwerpunktpraxis, Hanover
  - MediProjekt GbR, Hanover
  - Gemeinschaftspraxis Dr. Haytham Kamal und Dr. David C. Dorn, Hanover
  - Onkologische Schwerpunktpraxis, Heidelberg
  - SLK Kliniken Heilbronn Klinik für Innere Medizin III, Heilbronn
  - Cancer Center Zweiseenland GbR, Herrsching am Ammersee
  - Onkologische Schwerpunktpraxis im Medicinum, Hildesheim
  - Onkologische Schwerpunktpraxis Dres. Hansen & Reeb, Kaiserslautern
  - Klinikum Kassel, Klinik für Onkologie und Hämatologie, Kassel
  - Internisten am Markt, Köthen
  - MVZ Hämatologie und Onkologie Dr. Michael Neise & Dr. André Lollert, Krefeld
  - ÜBAG - MVZ Dr. Vehling-Kaiser GmbH, Landshut
  - Gemeinschaftspraxis für Hämatologie und Onkologie GbR, Lebach
  - Onkologie UnterEms Leer-Emden-Papenburg, Leer
  - MVZ Mitte am Johannisplatz, Leipzig
  - Mannheimer Onkologie Praxis, Mannheim
  - Gemeinschaftspraxis für Hämatologie & Onkologie, Moers
  - Brustzentrum Niederrhein im evangelischen Krankenhaus Bethesda, Mönchengladbach
  - Praxis für Hämatologie, Onkologie & Palliativmedizin, Mönchengladbach
  - MVZ Onkologie GmbH am Elisabeth-Krankenhaus Rheydt, Mönchengladbach
  - Gemeinschaftspraxis für Hämatologie internistische Onkologie, Mülheim
  - Medizinisches Zentrum für Hämatologie und Onkologie, München
  - Hämatologisch-onkologische Gemeinschaftspraxis, Münster
  - Friedrich-Ebert-Krankenhaus, Neumünster
  - TZN - Tumorzentrum Niederrhein GmbH, Neuss
  - MVZ Onko Medical GmbH Neustadt Innere, Med./Hämatologie-Onkologie, Neustadt am Rübenberge
  - Internistische Praxis und Tagesklinik, Neustadt i.S.
  - Onkologie Offenburg Ambulantes Therapiezentrum für Hämatologie und Onkologie, Offenburg
  - Pius-Hospital Oldenburg Hämatologie, Onkologie, Oldenburg
  - Onkologische Praxis Passau, Passau
  - Zentrum für Hämatologie und Onkologie MVZ GmbH, Porta Westfalica
  - MVZ für Blut- und Krebserkrankungen, Potsdam
  - Dr. Arnd Nusch, Ratingen
  - Studienzentrum Onkologie Ravensburg, Ravensburg
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Recklinghausen
  - Schwerpunktpraxis und Tagesklinik für Hämatologie und Onkologie, Regensburg
  - Praxis und Tagesklinik für Onkologie und Hämatologie, Remscheid
  - Onkologische Praxis Remscheid, Remscheid
  - Schwerpunktpraxis im Ärztehaus Rheinbach, Rheinbach
  - Gemeinschaftspraxis für internistische Hämatologie und Onkologie, Rheine
  - Praxis für Hämatologie und Internistische Onkologie, Rostock
  - Klinikum Südstadt Rostock Innere Medizin III, Rostock
  - GPR Gesundheits- und Pflegezentrum Rüsselsheim, Rüsselsheim am Main
  - Zentrum Ambulante Onkologie, Schorndorf
  - Schwerpunktpraxis für Hämatologie und Internistische Onkologie, Gastroenterologie, Singen (Hohentwiel)
  - MVZ Kloster Paradiese GbR, Soest
  - Hämatologie - Onkologie - Stolberg, Stolberg
  - Klinikum Stuttgart; Katharinenhospital Hämatologie, Onkologie und Palliativmedizin, Stuttgart
  - MVZ Leuschnerstr., Stuttgart
  - Kliniken Südostbayern - Klinikum Traunstein, Traunstein
  - Praxisnetzwerk Hämatologie / internistische Onkologie, Troisdorf
  - Onkologie Schwarzwald-Alb Dr. med. G. Köchling, Villingen-Schwenningen
  - Praxen MVZ für Innere Medizin, Weinheim
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Westerstede
  - Praxisgemeinschaft für Onkologie und Urologie, Wilhelmshaven
  - Internistische Gemeinschaftspraxis,Hämatologie, Onkologie,Palliativmedizin, Worms
  - MVZ West GmbH Würselen Hämatologie-Onkologie, Würselen
  - Hämatologisch-Onkologische, Schwerpunktpraxis Würzburg GbR,Dres. med. R. Schlag & B. Schöttker, Würzburg
  - Praxis und Tagesklinik für Hämatologie/Onkologie, Zittau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martens UM, Schroder J, Bengsch F, Sellmann L, Busies S, Frank-Gleich S, Zaiss M, Decker T, Schneeweiss A, Schuler M, Grebhardt S, Zacharias S, Marschner N, Kasenda B, Potthoff K, Vannier C. The INFINITY study protocol: a retrospective cohort study on decision making and clinical impact of biomarker-driven precision oncology in routine clinical practice. BMC Cancer. 2023 Jun 13;23(1):543. doi: 10.1186/s12885-023-11046-3. PMID 37312086